CLINICAL TRIAL: NCT02330692
Title: Cohort Study of New Prognostic Factors With Peripheral Blood and Bone Marrow Evaluation at the Time of Diagnosis and Relapse in Myelodysplastic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0479
Record Dates: First submitted 2014-12-25; First posted 2015-01-05 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Acquisition and storage of blood and bone marrow samples at diagnosis, at response evaluation and at times of relapse or refractory period.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Developing a molecular genetic test that can identify prognostic factors which can predict response to treatment, and to contribute to the establishment of future therapeutic strategies base on prognostic factors by undergoing peripheral blood and bone marrow examination of Myelodysplastic Syndrome (MDS) patients at diagnosis and relapse.

ELIGIBILITY:
Inclusion Criteria:

* MDS diagnosed by bone marrow aspiration and biopsy at Severance Hospital.

  * Male and Female over 16 years of age. ③ Written consent of the patient to participate in the cohort ④ Deaths during the study period are waiver of consent

Exclusion Criteria:

① Refusal or trouble understanding the written consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed with MDS in Severance Hospital. All patients are eligible for study occuring from the starting day of the study. Patients are enrolled if the written consent are acquired. Considering the annual incidence rate of the disease, target patient population is 1,000 people during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-09; Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
the number of patients with MDS to examine new prognostic factors | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea